CLINICAL TRIAL: NCT04372368
Title: Convalescent Plasma for the Treatment of Patients With COVID-19
Status: No longer available | Type: Expanded Access
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0990
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: COVID-19; SARS-CoV 2
Keywords: COVID-19; SARS-CoV-2; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: COVID-19 Convalescent Plasma — 1-2 units of COVID-19 convalescent plasma will be administered over 1 to 2 hours (rate of 100 to 200 mL/hr)

SUMMARY:
This expanded access program will provide access to COVID-19 convalescent plasma 150 or more individuals with moderate to severe or life-threatening manifestations of COVID-19, or documented to be at high risk of developing such manifestations at participating hospitals in Colorado.COVID-19 convalescent plasma is the liquid part of blood that is collected from patients who have recovered from COVID-19.

Convalescent plasma collected from individuals who have recovered from COVID-19 contains antibodies to SARS-CoV-2. Preliminary evidence and data collected during other respiratory virus outbreaks (including the 2003 SARS-CoV-1 epidemic, the 2009-2010 H1N1 influenza virus pandemic, and the 2012 MERS-CoV epidemic) suggest that the antibodies in convalescent plasma may be effective in fighting the infection.

DETAILED DESCRIPTION:
COVID-19 convalescent plasma will be obtained from FDA registered blood banks and will meet all regulatory requirements for conventional plasma and FDA's additional considerations for COVID-19 convalescent plasma (https://www.fda.gov/vaccines-blood-biologics/investigational-new-drug-ind-or-device-exemption-ide-process-cber/investigational-covid-19-convalescent-plasma-emergency-inds).

The primary objective of this expanded access program is to provide COVID-19 convalescent plasma to patients with moderate to severe or life-threatening manifestations of COVID-19, or documented to be at high risk of developing such manifestations.

The secondary objective will be the evaluation of safety, as assessed by incidents of adverse events judged by the treating physician to be potentially related to the administration of COVID-19 convalescent plasma.

Exploratory objectives will include assessments for antibody responses for patients that receive convalescent plasma. An exploratory analysis may be conducted correlating the level of neutralizing antibody titers with clinical outcomes observed. Due to the need to monitoring COVID19 antibody responses following infusion, blood testing at day 1 post-treatment and at discharge will be obtained as part of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed diagnosis of infection with SARS-CoV-2
* Age at least 18 years
* Laboratory confirmed diagnosis of infection with SARS-CoV-2
* Admitted to participating facility for the treatment of COVID-19 complications
* Moderate-to-Severe or life threatening COVID-19, or judged by the treating provider to be at high risk of progression to severe or life-threatening disease
* Informed consent provided by the patient or healthcare proxy
* Moderate COVID-19 is defined by one or more of the following:

  * Hospitalized with COVID-19
  * Respiratory rate >25/min
  * Oxygen saturation <96%
  * With or without radiographic evidence of pulmonary involvement
* Severe COVID-19 is defined by one or more of the following:

  * dyspnea
  * respiratory frequency ≥ 30/min
  * blood oxygen saturation ≤ 93%
  * Radiographic evidence of pulmonary disease
* Life-threatening COVID-19 is defined as one or more of the following:

  * respiratory failure requiring mechanical ventilation or non-rebreather oxygenation in the Intensive Care Unit.
  * Prone oxygenation.
  * multiple organ dysfunction or failure

Exclusion Criteria:

* Does not meet inclusion criteria
* History of transfusion reactions or contraindication to receiving convalescent plasma
* Risk of transfusion exceeds potential benefit based on clinician or blood bank determination.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: John D Beckham, MD, Principal Investigator — University of Colorado Denver, Anschutz Medical Campus
Locations (6):
- United States (6):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital North, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - UCHealth Poudre Valley Hospital, Fort Collins, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado